CLINICAL TRIAL: NCT02697162
Title: Antiseptic-coated Intermittent Urinary Catheter: Efficacy and Feasibility of Neurogenic Bladder Management and Prevention of Catheter-associated Urinary Tract Infections in Children
Brief Title: Antiseptic-coated Intermittent Urinary Catheter
Acronym: GuardianCath
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Withdrawal of research institution from participating
Sponsor: Children's Hospital Zagreb (Other)
Collaborators: GuardianMed j.d.o.o. Research and development in medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GCath-CHZ-01
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Neurogenic Bladder; Catheter-Related Infections
Keywords: Intermittent catheterisation; Antiseptic; Octenidine chloride; Children
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Catheter-Related Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antiseptic-coated catheter (Experimental): Hydrophilic intermittent urinary catheter coated with octenidine chloride
  Interventions: Device: Antiseptic-coated catheter; Drug: Octenidine chloride
- Hydrophilic catheter (Placebo Comparator): Hydrophilic intermittent urinary catheter
  Interventions: Device: Hydrophilic catheter

INTERVENTIONS:
Device: Antiseptic-coated catheter — Antiseptic-coated hydrophilic intermittent urinary catheter with octenidine chloride
  Other Names: GuardianCath
  Arms: Antiseptic-coated catheter
Device: Hydrophilic catheter — Hydrophilic intermittent urinary catheter
  Arms: Hydrophilic catheter
Drug: Octenidine chloride — Antiseptic
  Arms: Antiseptic-coated catheter

SUMMARY:
Study design is a prospective, randomised, double-blind, and interventional. Primary aim of the study is to investigate efficacy of antiseptic-coated intermittent hydrophilic urinary catheters in prevention and reduction of catheter-associated urinary tract infections in children with neurogenic bladder. Secondary aim is to assess feasibility of antiseptic-coated intermittent hydrophilic urinary catheters in neurogenic bladder management. Octenidine chloride will be used as antiseptic.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic bladder
* use of intermittent catheterisation for neurogenic bladder management
* informed oral and written consent from the child and both parents/legal guardian

Exclusion Criteria:

* Congenital anomalies of urinary tract or genitals
* Immunodeficiency
* Urinary tract fistula

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of urinary tract infections | 6 months after start of intervention
  Urinary tract infection is diagnosed when both urinalysis results disclose pyuria and/or bacteriuria and the presence of at least 1000 colony-forming units per mL of a uropathogen cultured from a urine specimen obtained through catheterization

SECONDARY OUTCOMES:
Safety during catheterisation | 6 months after start of intervention
  Discomfort during catheterisation will be measured by subjective evaluation on a 10-cm visual analogue scale (VAS), where 0 is 'no discomfort' and 10 is 'worst discomfort imaginable'. Pain, stinging, or resistance will be measured on a four-point scale (for example for pain: 1=no pain; 4=severe pain).
Adverse reactions | 6 months after start of intervention
  Adverse events (AEs) and serious AEs will be recorded by the investigator. The presence of visible bleeding will reported by the participants.
Expenses of infection-associated treatment | 6 months after start of intervention
  Total expenses in diagnostics and treatment of urinary tract infections
Improvement in health-related quality of life measured by PedsQL 4.0 Generic Core questionnaire | 6 months after start of intervention
  Improvement is defined by increase in total and subscale scores by more than defined minimally clinical important difference for PedsQL 4.0 Generic Core questionnaire

OTHER OUTCOMES:
Gut flora and catheter-associated infections | 2 years after start of intervention
  Impact of gut flora composition on incidence of catheter-associated urinary tract infections

CONTACTS AND LOCATIONS:
Overall Officials: Slaven Abdovic, MD, PhD, Principal Investigator — Children's Hospital Zagreb
Locations (1):
- Children's Hospital Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided